CLINICAL TRIAL: NCT07151157
Title: Therapeutic Value of Sirolimus in Refractory Adult-Onset Still's Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-495
Record Dates: First submitted 2025-08-24; First posted 2025-09-03 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-08

CONDITIONS: Adult-Onset Still's Disease
Keywords: Adult-Onset Still's disease; sirolimus; mTOR; ZFP36L2
MeSH Terms: conditions — Still's Disease, Adult-Onset

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sirolimus combination therapy group (Experimental): On the basis of the existing treatment, oral sirolimus will be added at a dose of two capsules per day, one in the morning and one in the evening.
  Interventions: Drug: add-on sirolimus therapy

INTERVENTIONS:
Drug: add-on sirolimus therapy — On the basis of the existing treatment, oral sirolimus will be added at a dose of two capsules per day, one in the morning and one in the evening.

SUMMARY:
This study aims to further evaluate the anti-inflammatory effects of the mTOR inhibitor sirolimus in patients with adult-onset Still's disease (AOSD), and to verify whether it can reduce inflammation and control disease activity by restoring ZFP36L2 expression and promoting the degradation of inflammatory cytokine mRNAs. A total of three patients with refractory AOSD will be enrolled, defined as those showing no significant improvement after treatment with glucocorticoids at 1 mg/kg, or experiencing relapse during tapering of glucocorticoids to 15 mg/day. On the basis of their existing therapy, patients will receive oral sirolimus at a dose of two capsules per day, one in the morning and one in the evening. On the day prior to initiating sirolimus and at weeks 4, 8, and 12 of treatment, 10 ml of peripheral blood will be collected by trained medical staff, and neutrophils will be isolated within 2 hours to assess ZFP36L2 expression levels. Throughout treatment, patients' clinical manifestations, including fever, rash, and joint pain, will be monitored, and dynamic changes in multiple inflammation-related markers will be measured in peripheral blood at weeks 4, 8, and 12. These include C-reactive protein (CRP), erythrocyte sedimentation rate (ESR), serum ferritin, soluble interleukin-2 receptor (sIL-2R), and a panel of cytokines. Finally, correlations among sirolimus treatment, ZFP36L2 expression, inflammatory responses, and disease activity will be analyzed to explore its potential therapeutic mechanisms in AOSD.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years;
2. Meeting the Yamaguchi criteria, with infection and malignancy excluded;
3. Meeting the definition of refractory AOSD, i.e., patients whose symptoms show no significant improvement after treatment with glucocorticoids at 1 mg/kg, or who experience relapse during tapering of glucocorticoids to 15 mg/d;
4. Complete clinical information;
5. Signed and dated informed consent form;
6. Willingness to comply with study procedures and cooperate throughout the entire study.

Exclusion Criteria:

1. Presence of other rheumatic diseases;
2. History of, or planned, hematopoietic stem cell transplantation;
3. Presence of severe comorbidities considered by the investigator to be unsuitable for participation in this clinical study, such as severe cardiac or pulmonary insufficiency, severe bone marrow suppression, or severe hepatic or renal dysfunction;
4. Acute conditions such as bowel perforation or complete intestinal obstruction;
5. Pregnant, planning pregnancy, or breastfeeding women;
6. Poor compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2025-08-30 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
AOSD Disease Activity Score | at weeks 12
  Pouchot Systemic Score Scoring items (1 point each): fever; arthritis/arthralgia; rash; sore throat; hepatosplenomegaly; pericarditis/pleuritis; lymphadenopathy; abnormal liver function; leukocytosis; hyperamylasemia/thrombocytopenia; elevated ESR or CRP; other systemic manifestations (e.g., myalgia, fatigue). Total score: 0-12 points, with higher scores indicating greater disease activity.

SECONDARY OUTCOMES:
AOSD Disease Activity Score | Baseline (day before sirolimus) and at weeks 4, and 8
  Pouchot Systemic Score Scoring items (1 point each): fever; arthritis/arthralgia; rash; sore throat; hepatosplenomegaly; pericarditis/pleuritis; lymphadenopathy; abnormal liver function; leukocytosis; hyperamylasemia/thrombocytopenia; elevated ESR or CRP; other systemic manifestations (e.g., myalgia, fatigue). Total score: 0-12 points, with higher scores indicating greater disease activity.
Serum C-reactive Protein (CRP) Concentration | Baseline (day before sirolimus) and at weeks 4, 8, and 12
  CRP will be measured from peripheral blood samples as a marker of systemic inflammation.
Erythrocyte Sedimentation Rate (ESR) | Baseline (day before sirolimus) and at weeks 4, 8, and 12
  ESR will be assessed from peripheral blood samples to evaluate inflammatory activity.
Concentration of Serum Ferritin | Baseline (day before sirolimus) and at weeks 4, 8, and 12
  Ferritin will be measured from peripheral blood samples as an indicator of disease activity and inflammation.
Level of Soluble Interleukin-2 Receptor (sIL-2R) | Baseline (day before sirolimus) and at weeks 4, 8, and 12
  sIL-2R will be measured from peripheral blood samples as a marker of immune activation.
Concentration of Inflammatory Cytokines (e.g., IL-6, TNF-α) | Baseline (day before sirolimus) and at weeks 4, 8, and 12
  Multiple inflammatory cytokines will be measured from peripheral blood samples to evaluate systemic inflammatory status.
Number of participants with Clinical symptoms such as rash and arthralgia | Baseline (day before sirolimus) and at weeks 4, 8, and 12
  Changes in clinical symptoms such as rash and joint pain will be observed and recorded through physical examination.
Expression level of ZFP36L2 in neutrophils | Baseline (day before sirolimus) and at weeks 4, 8, and 12
  Collect 10 mL of peripheral blood from patients and isolate neutrophils within 2 hours to measure the expression level of ZFP36L2.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruiiin Hospital Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No